CLINICAL TRIAL: NCT03105492
Title: Pregnant Women s Views About the Ethics of Prenatal Whole Genome Sequencing
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917080; 17-HG-N080
Record Dates: First submitted 2017-04-07; First posted 2017-04-10 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Pregnant
Keywords: Prenatal Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Pregnant women: Women who are pregnant

SUMMARY:
Background:

Prenatal whole genome sequencing (PWGS) will give expecting parents large amounts of genetic data about their baby. This raises ethical concerns. Researchers want to find out if women want access to the kind of data PWGS provides. They want to know why and under what circumstances women would or would not want the data.

Objective:

To explore the views of pregnant women about possible use of PWGS. To find out whether they would want different categories of genetic data, and how they would use such findings.

Eligibility:

Women ages 18 and older who pregnant and speak English or Spanish

Design:

Participants will be recruited by their doctors.

Participants will take a survey about their views of PWGQ. They may take it online or on paper.

DETAILED DESCRIPTION:
The impending implementation of prenatal whole genome sequencing (PWGS) raises a host of ethical concerns given the massive amounts of genetic information that expecting parents will be able to learn about their baby. This project involves a cross-sectional quantitative survey of pregnant women to explore whether they want access to the kinds of information provided by PWGS, why and under what circumstances. The survey will address questions such as: What sorts of information do pregnant women want to know about their baby, and why? What, if anything, would they do with the information? What kind of guidance would pregnant women like from their medical team regarding fetal genetic testing? Given the range of practical and ethical challenges posed by PWGS, our data will inform practitioners approaches towards PWGS as the technology develops and becomes more widely available. It is imperative that government regulators and professional societies take into account the views of people directly affected by any policies that are created - including patients themselves - before crafting rules for whether, when and how to utilize PWGS.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must be 18 years of age
* Participants must be pregnant
* Participants must speak English or Spanish

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women.
Sampling Method: Non-Probability Sample
Enrollment: 553 (Actual)
Dates: Start 2017-06-15 (Actual); Primary Completion 2018-02-12 (Actual); Study Completion 2019-04-10 (Actual)

PRIMARY OUTCOMES:
Views of pregnant women | at baseline
  This study seeks to explore the views of pregnant women about the hypothetical utility of PWGS, whether they would want different categories of genetic information, and how they would anticipate using such findings.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E Berkman, J.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- INOVA Fairfax Hospital, Falls Church, Virginia, United States